CLINICAL TRIAL: NCT06421727
Title: Rehabilitation Of Balance Function In Patients With Persistent Postural Perceptual Dizziness: A Longitudinal Study
Brief Title: Rehabilitation Of Balance Function In Patients With Persistent Postural Perceptual Dizziness.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nada Mostafa Abdelhamid, Assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-01-06MD
Record Dates: First submitted 2024-04-20; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Persistent Postural Perceptual Dizziness
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: combined vestibular rehabilitation incorporating optokinetic stimulation and virtual reality exercises on persistent postural perceptual dizziness patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation by optokinetic stimulation and virtual reality exercises . (Other): combined vestibular rehabilitation incorporating optokinetic stimulation and virtual reality exercises (by device Virtual reality system(Meta Quest 2_Advanced All-In-One Virtual Reality Headset_ 128 GB)) on persistent postural perceptual dizziness patients.
  Interventions: Other: Rehabilitation by optokinetic stimulation and virtual reality exercises .

INTERVENTIONS:
Other: Rehabilitation by optokinetic stimulation and virtual reality exercises . — Rehabilitation by optokinetic stimulation and virtual reality exercises(by deviceVirtual reality system(Meta Quest 2_Advanced All-In-One Virtual Reality Headset_ 128 GB)).

SUMMARY:
Rehabilitation Of Balance Function In Patients With Persistent Postural Perceptual Dizziness: A longitudinal Study

DETAILED DESCRIPTION:
this study will be conducted to show the long term effect of combined vestibular rehabilitation incorporating optokinetic stimulation and virtual reality exercises on persistent postural perceptual dizziness patients.

Aim:1.Evaluate the balance control function in patients with persistent postural perceptual dizziness using computerized dynamic posturography.

2.To study effect of rehabilitation using optokinetic stimulation and virtual reality on persistent postural perceptual dizziness patients.

3.To follow up patients after the vestibular rehabilitation therapy to study the persistence of improvement" if any" in patients with persistent postural perceptual dizziness .

Type of the study : prospective cohort and longitudinal study. Sources of data : Audio-vestibular medicine unit , Sohag University Hospital. Study group : consists of 36 patients age ranged from 18-65 years suffering from symptoms of persistent postural perceptual vertigo.

All subjects will be submitted to:

A- Detailed medical history, full history of dizziness. B-Acoustic impedance test. C-Basic audiological evaluation. D- Vestibular assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age: from 18 years to 65 years old.
* Gender: males and females.
* Can withstand and willing to undergo repeated vestibular rehabilitation therapy .*No history of any disease required to give treatment that could affect results.

Exclusion Criteria:

* Neurological disorders, paresis, paralysis, motor disorder, ataxia, brain mass, multiple sclerosis and stroke with grade 4 muscle power or below.
* Otological disorders e.g. middle ear pathology (chronic suppurative otitis media, Tumor).
* Psychiatric disorders e.g. Schizophrenia and endogenous depression.
* Severely ill patients who would not tolerate vestibular rehabilitation therapy .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Rehabilitation Of Balance Function In Patients With Persistent Postural Perceptual Dizziness : A longitudinal Study | 2 years
  Improvement of dizziness measured by Computerized dynamic posturography:6 conditions, the maximum handicap score 0/6 and the minimum 6/6.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ahmed, Study Chair — Sohag University

IPD SHARING:
Plan to Share IPD: No